CLINICAL TRIAL: NCT02899156
Title: Effect of Flumazenil on Hypoactive Delirium in the ICU: A Double-Blind, Placebo-Controlled Pilot Study
Brief Title: Flumazenil for Hypoactive Delirium Secondary to Benzodiazepine Exposure
Acronym: FLYP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A planned interim analysis led to the trial being stopped early based on the observed size effect and power analysis.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 837421
Record Dates: First submitted 2016-07-27; First posted 2016-09-14 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Hypoactive Delirium
Keywords: delirium; flumazenil; hypoactive delirium; benzodiazepine; benzodiazepine antagonist; critical care
MeSH Terms: conditions — Delirium | interventions — Flumazenil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flumazenil Infusion (Active Comparator): The flumazenil continuous infusion is started at an initial dose of 0.1 mg/hr., and can be titrated up to a maximum of 0.3 mg/hr. Dose titrations may occur every 60 minutes to maintain RASS scores of 0 to +1. The maximum rate is 0.3 mg/hr.
  Interventions: Drug: Flumazenil
- Placebo Infusion (Placebo Comparator): The placebo continuous infusion is started at an initial dose of 0.1 mg/hr (2 ml/hr)., and can be titrated up to a maximum of 0.3 mg/hr. Dose titrations may occur every 60 minutes to maintain RASS scores of 0 to +1. The maximum rate is 0.3 mg/hr.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flumazenil
  Other Names: Romazicon
  Arms: Flumazenil Infusion
Drug: Placebo — 0.9% normal saline
  Arms: Placebo Infusion

SUMMARY:
Delirium within the intensive care unit (ICU) is associated with poor outcomes such as increased mortality, ICU and hospital length of stay (LOS), and time on mechanical ventilation. Benzodiazepine (BZD) exposure is an independent risk factor for development of delirium. Reversal of hypoactive delirium represents a potential opportunity for reducing duration of delirium and subsequent complications.

This is a single-center randomized, double-blind, placebo-controlled study of critically ill adult patients with benzodiazepine-associated hypoactive delirium. The hypothesis is that flumazenil continuous infusion may reverse hypoactive delirium associated with BZD exposure and thereby reduce duration of delirium and ICU LOS.

DETAILED DESCRIPTION:
Benzodiazepines are commonly used for discomfort, anxiety, agitation, and alcohol withdrawal syndrome (AWS) in the ICU. End organ dysfunction and extended exposure can increase the risk of complications associated with BZDs, which include increased ICU LOS, time on mechanical ventilation, and mortality.

Flumazenil as a 1, 4-imidazobenzodiazepine is a competitive antagonist for the benzodiazepine binding site with weak intrinsic or partial agonistic activity on the GABA receptor. Multiple studies have confirmed the safety and effectiveness of flumazenil for the reversal of sedation. Pilot studies have demonstrated safe reversal of over-sedation and statistically significant improvements in patient cooperation and time to extubation. The current standard for suspected BZD-associated hypoactive delirium is cessation of benzodiazepine administration and supportive care.

The role of continuous infusion flumazenil for rapid and sustained reversal of hypoactive delirium in the ICU has not been evaluated prospectively and therefore remains poorly defined.

ELIGIBILITY:
Inclusion Criteria:

* critically ill adults
* RASS score of -3 to 0 after receiving benzodiazepine therapy
* CAM-ICU positive
* no benzodiazepine therapy within the previous 12 hours

Exclusion Criteria:

1. contraindications to flumazenil including hypersensitivity
2. receipt of benzodiazepines for control of potentially life-threatening conditions (e.g., control of intracranial pressure or status epilepticus)
3. active seizure disorder or on current anti-convulsant therapy for history of seizure disorder. Seizures secondary to alcohol withdrawal will NOT be excluded.
4. history of traumatic brain injury complicated by seizures
5. acute episode (within prior 30 days) of severe traumatic brain injury
6. history of structural lesion (e.g. subarachnoid hemorrhage, cerebrovascular accident, intra-parenchymal hemorrhage) complicated by seizures
7. acute episode (within prior 14 days) of structural lesion (e.g. subarachnoid hemorrhage, cerebrovascular accident, intra-parenchymal hemorrhage)
8. brain tumor complicated by seizure
9. history of anoxic brain injury
10. third-degree burn with total body surface area (TBSA) burn greater than 20%
11. chronic benzodiazepine (clonazepam:lorazepam:diazepam approximately 4:8:40 mg per day) for 7 consecutive days with no taper
12. chronic delirium that is attributable to other causes
13. anticipated to transfer to lower level of care within 24 hours
14. admitted for polysubstance overdose as determined by initial drug toxicity screening
15. recent exposure (prior 7 days) to pro-convulsant medications (identified via medication list, medication reconciliation performed by PI/pharmacy medication reconciliation team, or urine drug screening)
16. children, incarcerated individuals, and pregnant women
17. unable to provide consent and the legally authorized representative is unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra J Schomer, PharmD, Principal Investigator — University of California, Davis; Jeremiah J Duby, PharmD, BCPS, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandharipande P, Shintani A, Peterson J, Pun BT, Wilkinson GR, Dittus RS, Bernard GR, Ely EW. Lorazepam is an independent risk factor for transitioning to delirium in intensive care unit patients. Anesthesiology. 2006 Jan;104(1):21-6. doi: 10.1097/00000542-200601000-00005. PMID 16394685
- [Background] Zaal IJ, Devlin JW, Hazelbag M, Klein Klouwenberg PM, van der Kooi AW, Ong DS, Cremer OL, Groenwold RH, Slooter AJ. Benzodiazepine-associated delirium in critically ill adults. Intensive Care Med. 2015 Dec;41(12):2130-7. doi: 10.1007/s00134-015-4063-z. Epub 2015 Sep 24. PMID 26404392
- [Background] Shehabi Y, Bellomo R, Reade MC, Bailey M, Bass F, Howe B, McArthur C, Seppelt IM, Webb S, Weisbrodt L; Sedation Practice in Intensive Care Evaluation (SPICE) Study Investigators; ANZICS Clinical Trials Group. Early intensive care sedation predicts long-term mortality in ventilated critically ill patients. Am J Respir Crit Care Med. 2012 Oct 15;186(8):724-31. doi: 10.1164/rccm.201203-0522OC. Epub 2012 Aug 2. PMID 22859526
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Patel SB, Poston JT, Pohlman A, Hall JB, Kress JP. Rapidly reversible, sedation-related delirium versus persistent delirium in the intensive care unit. Am J Respir Crit Care Med. 2014 Mar 15;189(6):658-65. doi: 10.1164/rccm.201310-1815OC. PMID 24423152
- [Background] Brogden RN, Goa KL. Flumazenil. A reappraisal of its pharmacological properties and therapeutic efficacy as a benzodiazepine antagonist. Drugs. 1991 Dec;42(6):1061-89. doi: 10.2165/00003495-199142060-00010. PMID 1724638
- [Background] Breheny FX. Reversal of midazolam sedation with flumazenil. Crit Care Med. 1992 Jun;20(6):736-9. doi: 10.1097/00003246-199206000-00006. PMID 1597024
- [Background] Pepperman ML. Double-blind study of the reversal of midazolam-induced sedation in the intensive care unit with flumazenil (Ro 15-1788): effect on weaning from ventilation. Anaesth Intensive Care. 1990 Feb;18(1):38-44. doi: 10.1177/0310057X9001800107. PMID 2110788
- [Background] Penninga EI, Graudal N, Ladekarl MB, Jurgens G. Adverse Events Associated with Flumazenil Treatment for the Management of Suspected Benzodiazepine Intoxication--A Systematic Review with Meta-Analyses of Randomised Trials. Basic Clin Pharmacol Toxicol. 2016 Jan;118(1):37-44. doi: 10.1111/bcpt.12434. Epub 2015 Jul 28. PMID 26096314
- [Background] Kreshak AA, Cantrell FL, Clark RF, Tomaszewski CA. A poison center's ten-year experience with flumazenil administration to acutely poisoned adults. J Emerg Med. 2012 Oct;43(4):677-82. doi: 10.1016/j.jemermed.2012.01.059. Epub 2012 Jul 4. PMID 22766408
- [Background] Moore PW, Donovan JW, Burkhart KK, Waskin JA, Hieger MA, Adkins AR, Wert Y, Haggerty DA, Rasimas JJ. Safety and efficacy of flumazenil for reversal of iatrogenic benzodiazepine-associated delirium toxicity during treatment of alcohol withdrawal, a retrospective review at one center. J Med Toxicol. 2014 Jun;10(2):126-32. doi: 10.1007/s13181-014-0391-6. PMID 24619543
- [Background] Bodenham A, Park GR. Reversal of prolonged sedation using flumazenil in critically ill patients. Anaesthesia. 1989 Jul;44(7):603-5. doi: 10.1111/j.1365-2044.1989.tb11455.x. PMID 2505628
- [Background] Spivey WH, Roberts JR, Derlet RW. A clinical trial of escalating doses of flumazenil for reversal of suspected benzodiazepine overdose in the emergency department. Ann Emerg Med. 1993 Dec;22(12):1813-21. doi: 10.1016/s0196-0644(05)80407-x. PMID 8239101
- [Background] Salluh JI, Wang H, Schneider EB, Nagaraja N, Yenokyan G, Damluji A, Serafim RB, Stevens RD. Outcome of delirium in critically ill patients: systematic review and meta-analysis. BMJ. 2015 Jun 3;350:h2538. doi: 10.1136/bmj.h2538. PMID 26041151
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Krewulak KD, Stelfox HT, Leigh JP, Ely EW, Fiest KM. Incidence and Prevalence of Delirium Subtypes in an Adult ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 Dec;46(12):2029-2035. doi: 10.1097/CCM.0000000000003402. PMID 30234569
- [Background] Avelino-Silva TJ, Campora F, Curiati JAE, Jacob-Filho W. Prognostic effects of delirium motor subtypes in hospitalized older adults: A prospective cohort study. PLoS One. 2018 Jan 30;13(1):e0191092. doi: 10.1371/journal.pone.0191092. eCollection 2018. PMID 29381733
- [Background] Girard TD, Exline MC, Carson SS, Hough CL, Rock P, Gong MN, Douglas IS, Malhotra A, Owens RL, Feinstein DJ, Khan B, Pisani MA, Hyzy RC, Schmidt GA, Schweickert WD, Hite RD, Bowton DL, Masica AL, Thompson JL, Chandrasekhar R, Pun BT, Strength C, Boehm LM, Jackson JC, Pandharipande PP, Brummel NE, Hughes CG, Patel MB, Stollings JL, Bernard GR, Dittus RS, Ely EW; MIND-USA Investigators. Haloperidol and Ziprasidone for Treatment of Delirium in Critical Illness. N Engl J Med. 2018 Dec 27;379(26):2506-2516. doi: 10.1056/NEJMoa1808217. Epub 2018 Oct 22. PMID 30346242
- [Background] Ely EW. The ABCDEF Bundle: Science and Philosophy of How ICU Liberation Serves Patients and Families. Crit Care Med. 2017 Feb;45(2):321-330. doi: 10.1097/CCM.0000000000002175. PMID 28098628
- [Background] Bassett R, Adams KM, Danesh V, Groat PM, Haugen A, Kiewel A, Small C, Van-Leuven M, Venus S, Ely EW. Rethinking critical care: decreasing sedation, increasing delirium monitoring, and increasing patient mobility. Jt Comm J Qual Patient Saf. 2015 Feb;41(2):62-74. doi: 10.1016/s1553-7250(15)41010-4. PMID 25976892
- [Background] Balas MC, Vasilevskis EE, Olsen KM, Schmid KK, Shostrom V, Cohen MZ, Peitz G, Gannon DE, Sisson J, Sullivan J, Stothert JC, Lazure J, Nuss SL, Jawa RS, Freihaut F, Ely EW, Burke WJ. Effectiveness and safety of the awakening and breathing coordination, delirium monitoring/management, and early exercise/mobility bundle. Crit Care Med. 2014 May;42(5):1024-36. doi: 10.1097/CCM.0000000000000129. PMID 24394627
- [Background] Barnes-Daly MA, Phillips G, Ely EW. Improving Hospital Survival and Reducing Brain Dysfunction at Seven California Community Hospitals: Implementing PAD Guidelines Via the ABCDEF Bundle in 6,064 Patients. Crit Care Med. 2017 Feb;45(2):171-178. doi: 10.1097/CCM.0000000000002149. PMID 27861180
- [Background] Trogrlic Z, van der Jagt M, Lingsma H, Gommers D, Ponssen HH, Schoonderbeek JFJ, Schreiner F, Verbrugge SJ, Duran S, Bakker J, Ista E. Improved Guideline Adherence and Reduced Brain Dysfunction After a Multicenter Multifaceted Implementation of ICU Delirium Guidelines in 3,930 Patients. Crit Care Med. 2019 Mar;47(3):419-427. doi: 10.1097/CCM.0000000000003596. PMID 30608279
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Hojer J, Baehrendtz S, Magnusson A, Gustafsson LL. A placebo-controlled trial of flumazenil given by continuous infusion in severe benzodiazepine overdosage. Acta Anaesthesiol Scand. 1991 Oct;35(7):584-90. doi: 10.1111/j.1399-6576.1991.tb03353.x. PMID 1686131
- [Background] Weinbroum A, Rudick V, Sorkine P, Nevo Y, Halpern P, Geller E, Niv D. Use of flumazenil in the treatment of drug overdose: a double-blind and open clinical study in 110 patients. Crit Care Med. 1996 Feb;24(2):199-206. doi: 10.1097/00003246-199602000-00004. PMID 8605789
- [Background] Chern CH, Chern TL, Wang LM, Hu SC, Deng JF, Lee CH. Continuous flumazenil infusion in preventing complications arising from severe benzodiazepine intoxication. Am J Emerg Med. 1998 May;16(3):238-41. doi: 10.1016/s0735-6757(98)90091-2. PMID 9596422
- [Background] Flumazenil [package insert]. San Francisco, CA, Genentech Inc, 2010
- [Background] Devlin JW, Roberts RJ, Fong JJ, Skrobik Y, Riker RR, Hill NS, Robbins T, Garpestad E. Efficacy and safety of quetiapine in critically ill patients with delirium: a prospective, multicenter, randomized, double-blind, placebo-controlled pilot study. Crit Care Med. 2010 Feb;38(2):419-27. doi: 10.1097/CCM.0b013e3181b9e302. PMID 19915454

RESULTS

PARTICIPANT FLOW:
Groups:
- Flumazenil Group: The flumazenil continuous infusion is started at an initial dose of 0.1 mg/hr., and can be titrated up to a maximum of 0.3 mg/hr. Dose titrations may occur every 60 minutes to maintain RASS scores of 0 to +1. The maximum rate is 0.3 mg/hr.
  Flumazenil
- Placebo Group: The placebo continuous infusion is started at an initial dose of 0.1 mg/hr (2 ml/hr)., and can be titrated up to a maximum of 0.3 mg/hr. Dose titrations may occur every 60 minutes to maintain RASS scores of 0 to +1. The maximum rate is 0.3 mg/hr.
  Placebo: 0.9% normal saline
Period: Overall Study
Arm/Group | Flumazenil Group | Placebo Group
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Flumazenil Infusion: The flumazenil continuous infusion is started at an initial dose of 0.1 mg/hr., and can be titrated up to a maximum of 0.3 mg/hr. Dose titrations may occur every 60 minutes to maintain RASS scores of 0 to +1. The maximum rate is 0.3 mg/hr.
  Flumazenil
- Total: Total of all reporting groups
Arm/Group | Flumazenil Infusion | Placebo Infusion | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7) | 59.4 (7.6) | 58.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22
Days in Hospital Prior to Enrollment [Mean (Standard Deviation); unit: days] | 8.5 (2.8) | 10.6 (7.5) | 9.5 (5.8)
Time Since Last Benzodiazepine [Mean (Standard Deviation); unit: hours] | 43 (23) | 55 (37.1) | 49 (31.5)
Lorazepam Equivalents [Median (Inter-Quartile Range); unit: milligrams] | 117 [85.8 to 476] | 110.3 [57 to 221] | 113.6 [68.6 to 284.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Delirium-free Days
Description: Defined by the number of days in the 14-day period after randomization that the patient was alive and not delirious (i.e. CAM-ICU negative). Zero delirium-free days will be observed for patients that die within the 14-day period.
Time Frame: up to 14 days after randomization
Population: One patient randomized to the flumazenil and one randomized to the placebo never received the study infusion. The patient in the flumazenil group died from a massive hemorrhage within 1 hour of infusion initiation, and it was deemed nonattributable to study infusion. Twenty patients were included in the final analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Flumazenil Group | Placebo Group
Number analyzed (Participants) | 10 | 10
days | 12.7 [7.2 to 13.2] | 9.2 [0 to 10.2]

2. Secondary Outcome: Number of Participants With Delirium Resolution
Description: defined by the proportion of patients who were delirium free at 14 days after randomization
Time Frame: up to 14 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Flumazenil Group | Placebo Group
Number analyzed (Participants) | 10 | 10
Participants | 9 | 7

3. Secondary Outcome: Intensive Care Unit Length of Stay
Description: length of time that the patient was admitted to an intensive care unit service during the hospital stay
Time Frame: duration of admission to the intensive care unit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Flumazenil Group | Placebo Group
Number analyzed (Participants) | 10 | 10
days | 7.8 (4.8) | 7 (6)

4. Secondary Outcome: Number of Mechanical Ventilator Free Days
Description: number of days within the first 28 days after enrollment that the patient was free from needing mechanical ventilation
Time Frame: up to 28 days after randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Flumazenil Group | Placebo Group
Number analyzed (Participants) | 10 | 10
days | 23.6 (4.4) | 24.9 (5)

5. Secondary Outcome: Occurrence of Agitation Requiring Use of Rescue Sedatives While on Study Infusion
Description: number of times that a RASS score of + 2 to +4 occurred that did not resolve with decreasing study infusion
Time Frame: up to 72 hours after the start of the infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Flumazenil Group | Placebo Group
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

6. Secondary Outcome: Average Duration of Study Infusion
Description: average duration of time patient was randomized to each infusion up to 72 hours
Time Frame: up to 72 hours after the start of the infusion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Flumazenil Group | Placebo Group
Number analyzed (Participants) | 10 | 10
hours | 54.8 (16.8) | 58.2 (23.5)

7. Secondary Outcome: Average Maximum Rate of Study Infusion
Description: average maximum rate (ml/hr) during the 72 hours after study infusion
Time Frame: up to 72 hours after the start of the infusion
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Flumazenil Group | Placebo Group
Number analyzed (Participants) | 10 | 10
milliliters per hour | 5 (2) | 5.2 (2)

ADVERSE EVENTS:
Time Frame: 72 hours while on study infusion
Arm/Group | Flumazenil Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
A planned interim analysis led to the trial being stopped early based on the observed size effect and power analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT02899156/Prot_SAP_000.pdf